CLINICAL TRIAL: NCT03306433
Title: Prevention of Enamel Demineralization in Fixed Appliance Orthodontic Patients Using UDMA-K18 Sealant to Prevent Microbial Attachment Compared to a UDMA Control and no Sealant, a Randomized Split Mouth Clinical Trial
Brief Title: Prevention of Enamel Demineralization by Use of K18-smooth Surface Sealant
Acronym: K18
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado School of Dental Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17-0633
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Dental Caries
Keywords: dental caries; white spot lesion; prevention; smooth surface sealant
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: prospective, paired randomized control trial for which treatment (no sealant, UDMA control, UDMA-K18 sealant) will be applied clinically and evaluated on extracted teeth in laboratory conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial design is triple-blinded. The manufacturer will deliver the blinded treatments in identical bottles labelled A and B, therefore, neither the patient nor the clinician will know which treatment is rendered to each tooth. However, the no sealant control will not be blinded. Blinding will continue to be present during the histological portion of the experiment as the assessors will not be aware of which sealant was used to treat each tooth. After a blinded assessment, blinds will be lifted when between-group analysis is performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- UDMA-K18 (Experimental): UDMA-K18 smooth surface sealant
  Interventions: Device: UDMA-K18 smooth surface sealant
- UDMA-control (Placebo Comparator): UDMA smooth surface sealant without K18
  Interventions: Device: UDMA-K18 smooth surface sealant
- Negative control (No Intervention): No intervention to provide baseline

INTERVENTIONS:
Device: UDMA-K18 smooth surface sealant — The K18 as part of the UDMA polymer network (UDMA-K18) is hypothesized to prevent microbial attachment to the surface.
  Other Names: UDMA-control
  Arms: UDMA-K18; UDMA-control

SUMMARY:
This study will evaluate effectiveness of a urethane dimethacrylate (UDMA)-quaternary ammonium methacrylate (K18) resin (UDMA-K18) smooth surface sealant to prevent biofilm attachment to tooth surfaces thereby eliminating the possibility for the tooth to be demineralized. The hypothesis is that UDMA-K18 containing smooth surface sealant will be more effective at reducing enamel demineralization than the UDMA control or no treatment.

DETAILED DESCRIPTION:
Esthetics is a motivating factor to seek orthodontic treatment. However, if oral hygiene is inadequate during fixed appliance wear, unsightly white spot lesions (WSL) may develop. WSLs are areas of enamel demineralization that develop due to microbial assault that manifest as white, chalky opacity on the enamel. Urethane dimethacrylate (UDMA) can be modified to produce an antimicrobial compound, UDMA-K18, that has been proven to decrease microbial attachment in-vitro. (Sticker 2016) The use of a UDMA-K18 containing sealant may help to eliminate the development of WSLs around orthodontic brackets.

This study will place experimental or control smooth surface resins on teeth that are scheduled to be extracted for orthodontic reasons. These teeth are typically bicuspids that are to be extracted to create room for the orthodontic movement of teeth. These teeth are usually not extracted at the advent of first orthodontic bracket bonding but are extracted about 30 days later. The design of this study is to place sealants on those teeth (or as control, no sealant) and evaluate the teeth after they have been extracted.

Design: The study is a prospective, paired randomized control trial for which treatment (no sealant, UDMA-control, or UDMA-K18 sealant) will be applied clinically and evaluated on extracted teeth in laboratory conditions.

Procedures: Before bonding, one premolar per patient will be assigned to a group. The group each premolar is assigned to will be determined by a randomized, computer generated program. The allocation will be concealed in an opaque envelope that will be opened at the time of initial bonding. If a fourth premolar is planned for extraction, a random selection of the treatments will be selected in a 1:1:1 ratio and this treatment will be applied to the fourth premolar.

At the time of initial bonding, the UDMA and UDMA-K18 sealant will be applied to the selected premolar following manufacturer instructions. Briefly, the clinician will isolate the teeth using the NOLA Dry Field System and excess saliva will be removed by drying the teeth with an air-water syringe. In the treatment group, 37 % Phosphoric Acid will be applied to the entire buccal surface for 30 seconds, rinsed, and dried. Next, the assigned sealant will be evenly applied to the entire buccal surface of the premolar and light cured. The sealant which is adhesive will be applied to the bracket pad and the bracket pad will be pushed to place, excess cement will be removed and light cured.

In the control group, 37 % Phosphoric Acid will be applied for 30 seconds strictly to the area where the bracket will be bonded on the buccal surface, rinsed, and dried. No sealant will be applied. The adhesive sealant will be applied to the bracket pad and the bracket pad will be pushed to place, excess cement will be removed and light cured. After 3-6 weeks, the patient will have their premolars extracted. After extraction they will be placed in a Tooth Storage Solution (25 % ethanol, 75 % water with the addition of saturated hydroxyapatite, 20 mg of NaN3, and 40 mg Thymol) that is antimicrobial and does not alter the tooth surface. These teeth will be collected by the investigators for histologic study.

The collected, extracted teeth will be sectioned using a water-cooled, Buhler slow speed diamond saw in three 2mm sections through the bracket base. A polarized light microscopy (PLM) digitized photograph of the cross-sectional sample will be analyzed to determine the depth of lesions, if present. The mineral density profile will be analyzed using contact micro radiography (TMR).

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic patients at the Department of Orthodontics Clinic, School of Dental Medicine, University of Colorado who agree to consent to this study.
* Orthodontic treatment plans that include fixed appliances from the second premolar to second premolar in both arches.
* Orthodontic treatment plans that include extractions of at least 3 bicuspids at about 1 month after bracket placement.
* The patient has adequate oral hygiene

Exclusion Criteria:

* Evidence of decalcification or restorations on any of the premolars planned for extraction prior to orthodontic treatment,
* Pregnant women (self reported)
* Any condition that contraindicates orthodontic treatment,
* Not willing to consent to the study.

Ages: 12 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifton Carey, PhD, Principal Investigator — Professor, Dir Translational Research, University of Colorado, School of Dental Medicine
Locations (1):
- University of Colorado, School of Dental Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The COMIRB approval and the consent forms specify that we cannot share PHI except as mandated by law. Therefore we do not intend to share any IPD to other researchers.

REFERENCES:
- [Background] Schmuck BD, Carey CM. Improved Contact X-Ray Microradiographic Method to Measure Mineral Density of Hard Dental Tissues. J Res Natl Inst Stand Technol. 2010 Apr 1;115(2):75-83. doi: 10.6028/jres.115.006. Print 2010 Mar-Apr. PMID 21546983
- [Background] Gong SQ, Niu LN, Kemp LK, Yiu CK, Ryou H, Qi YP, Blizzard JD, Nikonov S, Brackett MG, Messer RL, Wu CD, Mao J, Bryan Brister L, Rueggeberg FA, Arola DD, Pashley DH, Tay FR. Quaternary ammonium silane-functionalized, methacrylate resin composition with antimicrobial activities and self-repair potential. Acta Biomater. 2012 Sep;8(9):3270-82. doi: 10.1016/j.actbio.2012.05.031. Epub 2012 May 29. PMID 22659173
- [Background] Liu SY, Tonggu L, Niu LN, Gong SQ, Fan B, Wang L, Zhao JH, Huang C, Pashley DH, Tay FR. Antimicrobial activity of a quaternary ammonium methacryloxy silicate-containing acrylic resin: a randomised clinical trial. Sci Rep. 2016 Feb 23;6:21882. doi: 10.1038/srep21882. PMID 26903314
- [Background] Wefel JS, Harless JD. Comparison of artificial white spots by microradiography and polarized light microscopy. J Dent Res. 1984 Nov;63(11):1271-5. doi: 10.1177/00220345840630110301. PMID 6094633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in January 2018 and ended in October 2018. Participants were recruited from the patient pool at the University of Colorado School of Dental Medicine Department of Orthodontics. Eligible candidates were offered the opportunity to participate in the study.
Pre-assignment Details: Participants were enrolled into the study if they met the inclusion criteria of having a planned orthodontic therapy that required extraction of at least 2 teeth and that those teeth were free of demineralization and did not have restorations.
Groups:
- All Participants: Participants were enrolled into the study if they met the inclusion criteria of having a planned orthodontic therapy that required extraction of at least 2 teeth and that those teeth were free of demineralization and did not have restorations. Enrolled participants were assigned to receive up to all three treatments. There were 16 participant total. Treatments included:
  UDMA-K18 smooth surface sealant: The K18 as part of the UDMA polymer network (UDMA-K18) is hypothesized to prevent microbial attachment to the surface.
  The adhesive used to bond the orthodontic bracket to the tooth UDMA-K18 smooth surface sealant: The K18 as part of the UDMA polymer network (UDMA-K18) is hypothesized to prevent microbial attachment to the surface.
Period: Overall Study
Arm/Group | All Participants
Started | 16
UDMA-K18 | 12
Adhesive Control | 12
UDMA-control | 9
Completed | 9
Not Completed | 7
Not completed — Lost to Follow-up | 3
Not completed — Patient did not have teeth extracted | 1
Not completed — Teeth not sent to the lab or participant only had two teeth for extraction | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants were enrolled into the study if they met the inclusion criteria of having a planned orthodontic therapy that required extraction of at least 2 teeth and that those teeth were free of demineralization and did not have restorations. All 16 participants had all three treatments. Thus there were 16 participant total. Treatments included:
  UDMA-K18 smooth surface sealant: The K18 as part of the UDMA polymer network (UDMA-K18) is hypothesized to prevent microbial attachment to the surface.
  The adhesive used to bond the orthodontic bracket to the tooth UDMA-K18 smooth surface sealant: The K18 as part of the UDMA polymer network (UDMA-K18) is hypothesized to prevent microbial attachment to the surface.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] — Participant age was self reported. All groups had the same participants
  Years
    Age | 13.8 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Canary Score [Mean (Full Range); unit: Canary Numbers] — The Canary Caries Detection System determines mineral quality (related to loss of mineral from the tooth). The measure is in Canary Numbers where 0 is no mineral loss and 100 is severe mineral loss.
  Canary Numbers | 7 [0 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Change in Mineral Density Determined by the Canary Caries Detection System
Description: The mineral density immediately below the surface of the tooth will lower if left unprotected to some extent.
Time Frame: Visit Window: 3-4 weeks.
Population: In this split mouth (same mouth) design all participants receive all treatments.
Measure: Mean (Standard Deviation); unit: Canary Number
Groups:
- Adhesive Control: The adhesive used to bond the orthodontic bracket to the tooth
Arm/Group | UDMA-K18 | UDMA-control | Adhesive Control
Number analyzed (Participants) | 12 | 9 | 12
Canary Number | 23.424 (3.288) | 31.125 (4.275) | 35.563 (7.378)
Statistical Analysis 1: Comparison: UDMA-K18 vs Adhesive Control; Paired difference test within each participant; Test type: Equivalence — The null hypothesis is that there are no significant paired differences between the groups. The power calculation is based on the observed variation and number of participants; p = 0.0003, Paired difference test, 2 sided — Paired difference p value comparing UDMA-K18 vs Adhesive Control; Paired difference t-test = -12.139, Standard Deviation 7.101 — There are 12 participants (pairs) for this comparison
Statistical Analysis 2: Comparison: UDMA-K18 vs UDMA-control; Paired comparison; Test type: Equivalence — Null hypothesis was that there were no differences between the groups; p = 0.0063, Paired difference test, 2 sided — Paired differrnce between UDMA-K18 and UDMA control; Paired difference t-test = -7.412, Standard Deviation 6.049 — There are 9 participant pairs for this comparison

2. Secondary Outcome: White Spot Lesion (WSL) Index
Description: The WSL Index is from 0 (no lesion) to 4 (severe lesion)
Time Frame: Visit Window: 3-4 weeks.
Population: Split mouth design : All participants received all treatments
Measure: Median (Full Range); unit: White spot Index
Arm/Group | UDMA-K18 | UDMA-control | Adhesive Control
Number analyzed (Participants) | 12 | 9 | 12
White spot Index | 0 [0 to 2] | 2 [0 to 2] | 2 [1 to 3]
Statistical Analysis 1: Comparison: UDMA-K18 vs Adhesive Control; WSL Index is non-parametric; Test type: Equivalence — The Null hypothesis was that there would be no differences between the groups; p = 0.0033, Chi-squared; Chi Square on WSL Index frequency = 15.77
Statistical Analysis 2: Comparison: UDMA-K18 vs UDMA-control; Test type: Equivalence — The null hypothesis was that there would not be any differences between the groups; p = 0.1450, Chi-squared; Chi Square on WSL Index frequency = 6.8321

ADVERSE EVENTS:
Time Frame: 10 Months, January 2018 to October 2018
Description: Study participants were provided with a 24-hour hot line to call if they experienced any discomfort associated with the placement of the sealant or orthodontic bracket.
Arm/Group | UDMA-K18 | UDMA-control | Adhesive Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT03306433/Prot_SAP_000.pdf